CLINICAL TRIAL: NCT05478889
Title: Surgical and Oncological Outcome After Minimally Invasive and Open Pancreatoduodenectomy for Distal Cholangiocarcinoma: an International Propensity Score Cohort Study
Brief Title: Minimally Invasive Pancreatoduodenectomy for Distal Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Sponsor
Other Study IDs: FPoliambulanza
Record Dates: First submitted 2022-07-22; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Distal Cholangiocarcinoma
Keywords: Minimally invasive pancreatoduodenectomy; Whipple; Distal cholangiocarcinoma; Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally invasive pancreatoduodenectomy: Whipple or pylorus preserving pancreatoduodenectomy following minimally invasive approach (laparoscopic or robotic). Hybrid (hand assisted) precedures will be included in the minimally invasive cohort.
  Interventions: Procedure: Minimally invasive pancreatoduodenectomy
- Open pancreatoduodenectomy: Whipple or pylorus preserving pancreatoduodenectomy following open (laparotomy) approach.

INTERVENTIONS:
Procedure: Minimally invasive pancreatoduodenectomy — Whipple's procedure using minimally invasive (laparoscopic/robotic) techniques
  Groups: Minimally invasive pancreatoduodenectomy

SUMMARY:
Outcomes for minimally invasive and open pancreatoduodenectomy for distal cholangiocarcinoma have not been compared. This is an international multicenter propensity score matched cohort study including patients after MIPD or OPD for dCCA. Primary outcomes included overall survival (OS) and disease-free interval (DFI).

DETAILED DESCRIPTION:
This study is an international multicenter propensity score matched cohort study using the database of the International Study Group on non-pancreatic periAmpullary CAncer, the ISGACA consortium (www.isgaca.com), including all patients who underwent a pancreatoduodenectomy for non-pancreatic periampullary cancer. Data will be retrospectively collected. To minimize differences between groups, all the participating centers perform both OPD and MIPD and all centers meet the Miami guideline minimum volume of at least 20 MIPD per year. This study is approved by all the locals Ethical Committees (approval number from the promoting center, Comitato etico di Brescia, NP 5318 - 01.06.2022) and it will be performed according to the STrengthening the Reporting of OBservational studies in Epidemiology (STROBE guideline and checklist), and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion criteria:

* Adult patients
* Elective upfront curative MIPD or OPD between January 1, 2010 and December 31, 2021
* Pathological confirmed dCCA

Exclusion criteria:

* Neoadjuvant chemotherapy
* Palliative surgical procedures
* Intraoperative detection of unresectable disease (i.e., metastasis or locally advanced disease)
* Post-operative pathological diagnosis was other than dCCA (e.g., neuroendocrine tumor, polyposis adenoma)
* R2 positive resection margin
* Pregnancy
* Missing primary endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients after elective upfront curative MIPD or OPD between January 1, 2010 and December 31, 2021 with a pathological confirmed dCCA
Sampling Method: Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Overall survival and disease-free interval | 60 months
  Time-to-event data, months + occurrence of event (death or recurrence)

SECONDARY OUTCOMES:
Major morbidity | 30 days or in-hospital
  Clavien-Diendo 3b-5

CONTACTS AND LOCATIONS:
Overall Officials: Moh'd Abu Hilal, MD, PhD, Principal Investigator — Fondazione Poliambulanza
Locations (1):
- Fondazione Poliambulanza Istituto Ospedaliero, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request it would be possible to share data.